CLINICAL TRIAL: NCT00552812
Title: Coarctation Of the Aorta Stent Trial
Acronym: COAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard E. Ringel (Other)
Responsible Party: Sponsor-Investigator, Richard E. Ringel, MD, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060057
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Coarctation of the Aorta
Keywords: Aortic Coarctation; Heart Defects, Congenital; Stents; Heart Catheterization
MeSH Terms: conditions — Aortic Coarctation; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stent therapy of aortic coarctation (Experimental): Stenting of aortic coarctation
  Interventions: Device: Stent therapy of aortic coarctation

INTERVENTIONS:
Device: Stent therapy of aortic coarctation — Transcatheter delivery of a metallic stent to enlarge region of aortic narrowing caused by the coarctation.
  Other Names: Cheatham-Platinum Stent

SUMMARY:
The purpose of this study is to determine whether Cheatham Platinum bare metal stents are safe and effective in the treatment of native and recurrent aortic coarctation in selected children, adolescents and adults.

DETAILED DESCRIPTION:
The goals of this study are to provide information that will support labeling of both the CP bare metal and covered stents to treat native and recurrent aortic coarctation in selected children, adolescents and adults. The investigation will have two phases: Phase One will examine the safety and efficacy of the bare metal stent, and will collect information about the covered stent when used as rescue therapy for aortic injuries occurring during bare metal stent procedures.

The aims of the Phase One study are to assess the use of the CP bare metal stent to:

1. provide a reduction equivalent to surgery in arm-leg systolic cuff blood pressure gradient 12 months after dilation and stent implantation, in comparison to the pre-dilation gradient;
2. accomplish gradient relief with a shorter number of days in hospital than surgery;
3. accomplish gradient relief with a rate of occurrence of serious procedure-related adverse events occurring within 30 days of dilation that is equivalent to surgery; and
4. accomplish gradient relief with a rate of occurrence of post-procedural paradoxical hypertension that is lower than surgery.

ELIGIBILITY:
Inclusion Criteria:

* Native or recurrent aortic coarctation
* Weight greater than or equal to 35 kg
* Noninvasive, arm-leg cuff systolic blood pressure difference or catheter measured systolic coarctation gradient greater than or equal to 20 mmHg

Exclusion Criteria:

* Age > 60 years
* Connective tissue disorders, including Marfan syndrome and other genetic syndromes such as Turner syndrome and Noonan syndrome
* Inflammatory aortitis
* Bloodstream infection, including endocarditis
* Pregnancy
* Aortic aneurysm
* Prior stent placement
* Adults lacking capacity to consent
* Foster children and/or wards of the court

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Ringel, MD, Principal Investigator — Johns Hopkins University; Kathy Jenkins, MD, Principal Investigator — Harvard University
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data is confidential and is not shared.

REFERENCES:
- [Derived] Hu L, Sun Q, Tang L, Cai M, Qian W, Dou T, Wang H, Wu Y, Liu Y. Food Effect on the Pharmacokinetics of VC004, a Tropomyosin Receptor Kinase Inhibitor: A Randomized Crossover Trial in Healthy Chinese Subjects. Clin Drug Investig. 2024 Jan;44(1):79-85. doi: 10.1007/s40261-023-01334-y. Epub 2023 Dec 19. PMID 38112942
- [Derived] Holzer RJ, Gauvreau K, McEnaney K, Watanabe H, Ringel R. Long-Term Outcomes of the Coarctation of the Aorta Stent Trials. Circ Cardiovasc Interv. 2021 Jun;14(6):e010308. doi: 10.1161/CIRCINTERVENTIONS.120.010308. Epub 2021 May 27. PMID 34039015
- [Derived] Meadows J, Minahan M, McElhinney DB, McEnaney K, Ringel R; COAST Investigators*. Intermediate Outcomes in the Prospective, Multicenter Coarctation of the Aorta Stent Trial (COAST). Circulation. 2015 May 12;131(19):1656-64. doi: 10.1161/CIRCULATIONAHA.114.013937. Epub 2015 Apr 13. PMID 25869198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened February, 2008 and ended December, 2010
Pre-assignment Details: Patients were consented as outpatients, but final selection criteria were assessed in the catheterization laboratory
Groups:
- Coarctation Stenting: Stent enlargement of aortic coarctation : Transcatheter delivery of a metallic stent to enlarge region of aortic narrowing caused by the coarctation.
Period: Overall Study
Arm/Group | Coarctation Stenting
Started | 105 (168 consents, 57 failed cath criteria, 5 met criteria but received covered stent, 1 withdrew consent)
Completed | 85 (Some still remain inside the 2 year follow up window. 2 year follow up data is not yet complete.)
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Coarctation Stenting
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [8 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 73
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in Difference Between Arm and Leg Systolic Blood Pressure From Baseline to 12 Months
Description: Noninvasive systolic blood pressures are measured in the arms and legs at baseline and 12 month follow-up. The difference between these measurements are calculated. The difference between systolic arm and leg blood pressures decreased by 30 ± 22 mmHg (n=90)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Coarctation Stenting: Stent enlargement of aortic coarctation: Transcatheter delivery of a metallic stent to enlarge region of aortic narrowing caused by the coarctation.
Arm/Group | Coarctation Stenting
Number analyzed (Participants) | 90
mmHg | 30 (22)

2. Secondary Outcome: Percentage of Participants With a Systolic Blood Pressure Greater Than the 95th Percentile for Age and Gender 12 Months Post Stent Placement
Description: Noninvasive Blood pressure is assessed at baseline and 12 months. The number of patients with a Systolic Blood Pressure > 95th Percentile for Age and Gender is recorded at Baseline (n=105) and compared to 12 month follow up (n=92).
Time Frame: Baseline and 12 months
Population: Study patients compared at baseline and within the 12 month follow up window: Baseline (n=105) compared to 12 month follow up (n=92)
Measure: Number; unit: percentage of participants
Arm/Group | Coarctation Stenting
Number analyzed (Participants) | 105
percentage of participants
  Baseline | 61
  12 month follow up | 17

3. Secondary Outcome: Systolic Blood Pressure, Difference Between Upper and Lower Extremities
Description: Measurement of difference between upper and lower extremities by noninvasive, automated measurement of four quadrant Systolic Blood Pressure. Comparison between baseline and 12 month follow up.
Time Frame: Baseline and 12 months
Population: Comparison between baseline(n=105) and 12 month follow up (n=92)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Coarctation Stenting
Number analyzed (Participants) | 105
mmHg
  Baseline | 29 (17)
  12 months | -1 (15)

ADVERSE EVENTS:
Arm/Group | Coarctation Stenting
Serious Adverse Events (participants affected / at risk) | 1/105
Other Adverse Events (participants affected / at risk) | 14/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coarctation Stenting (N=105)
Abnormal exercise echo test at one year (Cardiac disorders) | 1 — Hypertension on exercise testing related to residual stent narrowing
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coarctation Stenting (N=105)
Localized vascular tear (Vascular disorders) | 2
Aortic Aneurysm (Cardiac disorders) | 5
Post-procedure hypertension (Cardiac disorders) | 2
Residual aortic obstruction (Cardiac disorders) | 2
Stent Malposition (Cardiac disorders) | 1
AV Fistula (Cardiac disorders) | 1
Groin Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No